CLINICAL TRIAL: NCT04122417
Title: The Effect Of Therapeutic Touch Training Given To Mothers With Preterm Babies On Attachment Level And The Responses The Baby
Brief Title: The Effect Of Therapeutic Touch To Mothers With Preterm Babies
Status: Completed | Type: Observational
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Seyda Can, Director, University of Yalova
Other Study IDs: YALOVA ÜNİVERSİTESİ
Record Dates: First submitted 2019-10-08; First posted 2019-10-10 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Therapeutic Touch
Keywords: Therapeutic touch; yakson; gentle human touch; maternal attachment; preterm baby

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group: The mothers and infants in the experimental and control groups were assigned to the groups by randomization method. Therapeutic touch didn't apllied to control group.
  Babies in the control group who took care practices in accordance with normal hospital procedures.
  Interventions: Other: The Effect Of Therapeutic Touch Training Given To Mothers With Preterm Babies On Attachment Level And The Responses The Baby
- Yakson Group: The touch method was taught to the mothers in the Yakson group by the researcher in the first three days after the birth with the training brochure, video and applications on the model that are prepared in accordance with expert opinion.
  In yakson method, mother's fingers are closed, and she should touch in a way that does not apply excessive pressure. The method is applied for a total of 15 minutes in three cycles. First 5 minutes is resting the hand, 5 minutes is gentle caressing, and another 5 minutes of resting the hand.
  Interventions: Other: The Effect Of Therapeutic Touch Training Given To Mothers With Preterm Babies On Attachment Level And The Responses The Baby
- Gentle Human Touch Group: The touch method was taught to the mothers in the Gentle Human Touch group by the researcher in the first three days after the birth with the training brochure, video and applications on the model that are prepared in accordance with expert opinion.
  Mother slowly places one hand on the baby's hand and the other over pelvic cavity, covering the waist and hips of the baby.
  The touch is preserved for 15 minutes. In order to ensure equal touch for the duration of gentle human touch, the mother sits on a stool and her elbows have to be at the same level with baby's bed
  Interventions: Other: The Effect Of Therapeutic Touch Training Given To Mothers With Preterm Babies On Attachment Level And The Responses The Baby

INTERVENTIONS:
Other: The Effect Of Therapeutic Touch Training Given To Mothers With Preterm Babies On Attachment Level And The Responses The Baby — The study was carried out as randomized experiment to determine the effect of Yakson or Gentle Human Touch method practiced by mothers to preterm newborns on the maternal attachment level and the baby's responses.
  Other Names: The Effect Of Yakson Or Gentle Human Touch

SUMMARY:
The study was carried to determine the effect of yakson or gentle human touch methods applied by the mothers to their preterm newborns on mother's attachment level and baby's response.

DETAILED DESCRIPTION:
The study was carried out as a randomized controlled experimental research. Population of the study is all of the babies who were hospitalized at the neonatal intensive care unit of a state hospital in Turkey between August 2016 and August 2017 and the mothers of the babies; its sample is 90 mothers and their babies included with randomization method who were matching the criteria who were also hospitalized between these dates.

ELIGIBILITY:
Inclusion Criteria:

Mothers' Selection Criteria

* Mother should not have any defines psychiatric diseases,
* Mother should not have any physical disabilities,
* Mother should be literate and open to communication,
* Should not have transportation problem,
* Should be willing to participate and volunteer for the study.

Babies' Selection Criteria

* Babies should be between 26-34 gestation weeks,
* Should not have congenital abnormalities,
* Babies should not have any health problems that may hinder the practice (Intracranial hemorrhage, sepsis, hemorrhagic diseases, having an operation, etc.).

Exclusion Criteria:

-Participants must have inclusion criterias.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The sample of the study consists of babies and their mothers who were matching the criteria of the research between these dates and who volunteered. As a result of the power analysis, sample size was calculated as 90 for experimental and control groups with Power: 0.80. As a result of the sample calculation a total of 90 mothers and babies; 30 for Yakson group, 30 for gentle human touch group, 30 for control group were included in the study. The assignment of mothers and babies to the experiment and control groups was carried out by randomization with drawing lots method.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
The Effect Of Therapeutic Touch Training Given To Mothers With Preterm Babies On Attachment Level And The Responses The Baby | Between August 2016 and August 2017
  Study was determined that therapeutic touch methods applied to babies by the mothers increase mother-baby attachment; contributed to the sleep-calmness states, vital signs and weight gain of the baby; and reduced the stays in hospital.

CONTACTS AND LOCATIONS:
Overall Officials: ŞEYDA CAN, PhD, Principal Investigator — university

IPD SHARING:
Plan to Share IPD: No